CLINICAL TRIAL: NCT04915183
Title: Phase II Interventional Study Using Atorvastatin to Reduce Cisplatin-Induced Hearing Loss Among Individuals With Head and Neck Cancer
Brief Title: Atorvastatin to Reduce Cisplatin-Induced Hearing Loss Among Individuals With Head and Neck Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 210002; 21-DC-0002
Record Dates: First submitted 2021-06-04; First posted 2021-06-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Hearing Loss; Head and Neck Cancer
Keywords: Audiogram; Statin; Chemotherapy; Squamous Cell Carcinoma
MeSH Terms: conditions — Hearing Loss; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Atorvasatatin (40 mg)
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo will be formulated to also contain a white powder such that the atorvastatin and placebo are indistinguishable even if a capsule is opened.
  Arms: 2
Drug: Atorvastatin — Subjects will be provided with atorvastatin (40 mg) or placebo to be taken daily by mouth or by feeding tube. The tablets may be taken whole or crushed according to patient swallowing capabilities and preference.
  Arms: 1

SUMMARY:
Background:

Cisplatin is used to treat head and neck cancer. People who take this drug are at risk for hearing loss. Atorvastatin is a drug used to treat high cholesterol. It might reduce the risk of cisplatin-induced hearing loss.

Objective:

To find out if atorvastatin reduces hearing loss in people treated with cisplatin and radiation.

Eligibility:

People ages 18 and older with squamous cell carcinoma of the head and neck who will undergo treatment with cisplatin-based chemotherapy and radiation

Design:

Participants will be screened with their medical records.

Participants currently taking a cholesterol-lowering statin medication are invited to participate in the observational arm of the study. Those not taking such a medication are invited to participate in the interventional arm of the study.

All participants will have 3 study visits for the purpose of evaluating hearing. One before starting cisplatin treatment, one within 3 months of completing cancer treatment, and one within 2 years of completing cancer treatment. They will have tympanograms. A small flexible tip will be placed in the ear canal. A puff of air will be delivered to assess mobility of the ear drum. They will have hearing tests. They will wear headphones. They will listen to tones that vary in loudness. They will be asked to indicate when they hear a sound. They will complete 3 questionnaires at the time of each hearing test.

Participants will have 2 visits for blood tests. These will occur upon consent and 12 weeks after. They will be randomly assigned to take the study drug or placebo orally, once daily. They will take it during cisplatin treatment and for 3 months after treatment.

Long-term follow up will include a chart review 2 years after participants complete their cisplatin therapy.

DETAILED DESCRIPTION:
Study Description: Individuals undergoing cisplatin-based chemotherapy are at risk for developing significant, permanent hearing loss. The cholesterol-lowering drug atorvastatin has the potential to reduce the incidence and severity of hearing loss, as evidenced by our preclinical data in mice and our retrospective data in humans. Here we will compare hearing changes between subjects on a concurrent 40 mg daily dose of atorvastatin vs. a placebo among individuals undergoing cisplatin-based chemotherapy to treat head and neck cancer.

Objectives:

Primary Objective: To determine the effectiveness of atorvastatin (40 mg) in subjects treated with cisplatin-based chemotherapy for head and neck squamous cell carcinoma (HNSCC) at reducing moderate changes in hearing sensitivity relative to baseline, as defined by CTCAEv5.0 Grade>=2 criteria.

Secondary Objectives:

* To determine disease-free survival and overall survival in subjects undergoing cisplatin-based chemotherapy.
* To determine whether atorvastatin increases grade 3-5 treatment emergent adverse events versus placebo
* To determine the effectiveness of atorvastatin (40 mg) at reducing changes in hearing sensitivity relative to baseline, as defined by ASHA criteria, in subjects treated with cisplatin- based chemotherapy for head and neck squamous cell carcinoma (HNSCC).

Endpoints:

Primary Endpoint: The incidence of hearing loss at 12 +/-4 weeks after completion of cisplatin-based chemotherapy). Hearing loss will be defined according to CTCAEv5.0 Grade >=2 criteria based on changes in sensitivity relative to baseline, in at least one ear, across 1, 2, 3, 4, 6 and 8 kHz and will be compared in subjects taking atorvastatin (40 mg) vs. subjects taking placebo.

Secondary Endpoints:

* Overall and disease-free survival at 2 years after cisplatin-based chemotherapy. Overall survival and disease-free median survival will be compared between subjects taking atorvastatin (40 mg) vs. those taking placebo.
* Incidence of new CTCAEv5.0 grade > 3 AEs through 12 weeks after chemotherapy in the placebo and atorvastatin arms.
* Incidence of hearing loss at 12 +/- 4 weeks after completion of cisplatin-based chemotherapy. Hearing loss will be defined according to ASHA criteria based on changes in sensitivity relative to baseline, in at least one ear, across 1, 2, 3, 4, 6, 8, 10, and 12.5 kHz and will be compared in subjects taking atorvastatin (40 mg) vs. subjects taking placebo.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria evaluated by the study team, including an on-site oncologist:

* Willingness and ability to comply with and participate in all study procedures and availability for the duration of the study
* Ability to provide consent and provision of signed and dated informed consent form
* Adult subjects, aged >=18
* Diagnosed with squamous cell carcinoma of the head and neck, confirmed by a pathologic review of surgical or biopsy specimen(s), who meet standard clinical and laboratory criteria and will undergo treatment with concomitant cisplatin-based chemotherapy and radiation with curative intent or treatment with neoadjuvant chemotherapy (NAC). This includes subjects who will be treated with either intensity-modulated radiation therapy (IMRT) or proton radiotherapy, with planned dose to the cochlea <35 Gy (to limit confounding effects of radiation). Patients receiving immunotherapy in addition to cisplatin chemoradiation are eligible. Subjects treated with either high-dose cisplatin (typically 100 mg/m^2 x 2-3 doses every three weeks) or low-dose, weekly cisplatin (typically 40 mg/m^2 x 6-7 doses weekly) may enroll. Cisplatin in the neo-adjuvant setting may be given within a combination chemotherapy regimen (e.g TPF= Docetaxel, Cisplatin and 5FU or DC = Docetaxel Cisplatin)
* Subjects must have hearing thresholds at or better than 70 dB HL at 1, 2, and 4 kHz in at least one ear at the time of their baseline audiogram. CTCAE criteria (primary endpoint) and ASHA criteria (secondary endpoint) are based on changes in hearing in at

least one ear with one ototoxicity event/grade assigned per person.

* Baseline laboratory tests with lab values <1.5x the upper limit of normal: aspartate aminotransferase (AST or SGOT); alanine aminotransferase; creatine phosphokinase, creatinine
* Ability to take oral medication by mouth or by feeding tube and willingness to adhere to the daily atorvastatin or placebo regimen
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to enrollment and agreement to use such a method during study participation and for an additional 8 weeks after the end of atorvastatin administration

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Subjects currently taking a statin drug
* Subjects with bilateral flat, Type B tympanogram
* Subjects with bilateral cochlear implants
* Pre-existing liver or kidney disease that in the opinion of the investigator would interfere with taking Atorvastatin 40 mg daily.
* Subjects with a history of prior treatment with platinum chemotherapy drugs
* Staff members of the NIDCD Sections and of the lead site investigators headed by the PIs
* Children will be excluded because HNSCC in children under age 18 is exceedingly rare
* Current use of cimetidine, spironolactone, ketoconazole, cyclosporine, protease inhibitors, gemfibrozil, clarithromycin or itraconazole
* Pregnancy, lactation, or plan to become pregnant
* Known allergic reactions to components of atorvastatin or the placebo
* Other severe or unstable medical conditions which clinical site PI believes increase risk to safety or ability to complete study
* Expected concomitant use of aminoglycoside antibiotics

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of atorvastatin (20 mg) at reducing the incidence and severity of cisplatin-induced hearing loss in patients with head and neck squamous cell carcinoma (HNSCC). | Baseline (prior to treatment) to a repeated audiogram at the end of treatment (within 2-4 months of cessation of cisplatin administration).
  The primary endpoint is the change in hearing sensitivity (as measured by pure-tone audiometry) between the pre-treatment (before cisplatin therapy) hearing test and the post-treatment (after completion of cisplatin therapy) audiogram. Hearing loss will be defined according to CTCAE criteria and will be compared in subjects taking atorvastatin vs. subjects not taking any statin drug. Hearing sensitivity will be compared between audiograms collected at baseline (prior to treatment) to a repeated audiogram at the end of treatment (within 2-4 months of cessation of cisplatin administration).

SECONDARY OUTCOMES:
To examine the extent to which atorvastatin 40 mg alters overall survival and disease-free survival. | The overall survival and disease-free survival will be assessed at 3 months, 1 and 2 years after cisplatin-based CRT. Overall complete clinical response, comparing subjects taking atorvastatin (40 mg) vs those taking placebo.
  It is important to confirm that atorvastatin use does not reduce overall response, survival or disease- free survival in subjects with HNSCC. To date, only two retrospective studies have compared survival in HNSCC subjects taking statins.
To compare the incidence of grade (Bullet)3 AEs through 4 weeks after CRT with atorvastatin versus placebo. | Another secondary endpoint will be the incidence of grade (Bullet)3 AEs, which are expected to occur with CRT but rarely with atorvastatin.
  It is important to confirm that atorvastatin does not increase the overall toxicity associated with CRT.
To determine the effectiveness of atorvastatin (40 mg) at reducing changes in hearing sensitivity relative to baseline, as defined by ASHA criteria, in subjects treated with cisplatin- based CRT for head and neck squamous cell carcinoma (HNSCC). | The incidence of hearing loss at 12 4 weeks after completion of cisplatin-based CRT. Hearing loss will be defined according to ASHA criteria, comparing subjects taking atorvastatin (40 mg) vs. placebo.
  The American Speech-Langauge-Hearing Association (ASHA) ototoxicity criteria can be used for early detection based on changes in hearing sensitivity in extended high frequencies (>8 kHz). While ASHA does not assign grades to indicate severity, it may provide early diagnosis of hearing loss that has not yet spread to speech-related frequency regions of the cochlea (<8 kHz).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L Cunningham, Ph.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (4):
- United States (4):
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Wilmot Cancer Institute at the University of Rochester Medical Center in New Yor, Rochester, New York

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-DC-0002.html